CLINICAL TRIAL: NCT00110591
Title: A Phase I, Randomized, Double Blind, Placebo Controlled, Single-Dose, Rising Dose Cohort Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PRO 140 in Healthy Volunteers
Brief Title: Safety and Tolerability of PRO 140 in HIV Uninfected Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5R44AI046871-04 (NIH); PRO140-1101 (Other: CytoDyn)
Record Dates: First submitted 2005-05-10; First posted 2005-05-11 (Estimated); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Intravenous placebo for PRO 140
  Interventions: Drug: PRO 140
- PRO 140 dose 1 (Experimental): 0.1 mg/kg PRO 140 by intravenous infusion
  Interventions: Drug: PRO 140
- PRO 140 dose 2 (Experimental): 0.5 mg/kg PRO 140 by intravenous infusion
  Interventions: Drug: PRO 140
- PRO 140 dose 3 (Experimental): 2.0 mg/kg PRO 140 by intravenous infusion
  Interventions: Drug: PRO 140
- PRO 140 dose 4 (Experimental): 5.0 mg/kg PRO 140 by intravenous infusion
  Interventions: Drug: PRO 140

INTERVENTIONS:
Drug: PRO 140 — Monoclonal antibody to CCR5
  Other Names: Humanized monoclonal antibody to CCR5

SUMMARY:
The purpose of the study is to determine the safety and tolerability of PRO 140, an investigational anti-HIV drug, administered via intravenous infusion.

Study hypothesis: Single intravenous doses of PRO 140 can be safely administered to humans and will result in measurable concentrations of the product in serum.

DETAILED DESCRIPTION:
PRO 140 is a man-made monoclonal antibody to the chemokine receptor CCR5, which serves as a co-receptor for HIV. In numerous preclinical models of HIV infection, PRO 140 broadly and potently blocks CCR5-mediated HIV entry without blocking the natural activity of CCR5. PRO 140 is being developed for therapy of HIV infected individuals. The purpose of this study is to evaluate the safety and tolerability of PRO 140 in HIV uninfected male volunteers. The pharmacokinetics and pharmacodynamics of PRO 140 will also be assessed in this study.

Participants in this study will be randomly assigned to receive a single dose of one of several possible doses of PRO 140 or placebo. Participants will remain in the clinic for observation and evaluation for 24 hours after the single-dose administration. Follow-up visits will occur at 2, 3, 5, 7, 10, 14, 28, 42, and 60 days post-treatment. Physical exams, electrocardiograms (ECGs), vital signs measurement, adverse event reporting, and blood and urine collection will occur at most visits.

ELIGIBILITY:
Inclusion Criteria:

* Not more than 20% below or 20% above ideal weight for height and estimated frame size
* Good health, with no clinically significant abnormal findings on the physical examination, medical history, or laboratory tests

Exclusion Criteria:

* History of clinically significant disease
* History of clinically significant allergies, including drug allergy
* Participated in another clinical trial within the 3 months prior to study entry
* HIV infected
* Hepatitis B or C virus infected
* Active significant infection
* Prior exposure, allergy, or known hypersensitivity to PRO 140

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04-16; Primary Completion 2005-11-07 (Actual); Study Completion 2008-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Olson, PhD, Study Chair — Vice President, Clinical Research, Progenics Pharmaceuticals, Inc.
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | PRO 140 Dose 1 | PRO 140 Dose 2 | PRO 140 Dose 3 | PRO 140 Dose 4
Started | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PRO 140 Dose 1 | PRO 140 Dose 2 | PRO 140 Dose 3 | PRO 140 Dose 4 | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 4 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (7) | 34 (13) | 30 (12) | 22 (2) | 21 (2) | 27 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 4 | 4 | 20
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of PRO 140
Time Frame: 60 days
Measure: Number; unit: number of subjects reporting AEs
Arm/Group | Placebo | PRO 140 Dose 1 | PRO 140 Dose 2 | PRO 140 Dose 3 | PRO 140 Dose 4
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
number of subjects reporting AEs | 4 | 4 | 0 | 4 | 3

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over an 18-month period.
Description: Adverse events were systematically assessed through documented physical examinations, vital sign evaluation, ECGs as well as hematology, uranalysis and chemistry labs. All information is collected on case report forms.
Arm/Group | Placebo | PRO 140 Dose 1 | PRO 140 Dose 2 | PRO 140 Dose 3 | PRO 140 Dose 4
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 0/4 | 4/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | PRO 140 Dose 1 (N=4) | PRO 140 Dose 2 (N=4) | PRO 140 Dose 3 (N=4) | PRO 140 Dose 4 (N=4)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — 38 days after receiving PRO 140 (0.1 mg/kg) dose, subject suffered myocardial infarction. This was determined not related to study drug. Subject had severe atherosclerotic disease and history of chest pains.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | PRO 140 Dose 1 (N=4) | PRO 140 Dose 2 (N=4) | PRO 140 Dose 3 (N=4) | PRO 140 Dose 4 (N=4)
Fatal Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — This occurred 38 days after administration of the study drug at dose 0.1 mg/kg.
high creatine phosphokinase level (Investigations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (3) — one subject (5 mg/kg) had a severe grade 3 AE. There was a grade 3 increased creatine phosphokinase (CPK) test result.
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loose stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (6) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other